CLINICAL TRIAL: NCT06449235
Title: Efficacy and Safety of Omarigliptin, A Weekly Dipeptidyl Peptidase-4 Inhibitor for Type 2 Diabetes Management: Real-World Evaluation in Bangladesh
Brief Title: Real-World Evaluation of Omarigliptin for Type 2 Diabetes Meliitus in Bangladesh
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bangladesh Institute of Research and Rehabilitation in Diabetes, Endocrine and Metabolic Disorders (Other)
Collaborators: Pi Research and Development Center (Unknown); Acme Laboratories Ltd. (Unknown)
Responsible Party: Principal Investigator, Professor Dr. Feroz Amin, Head of the Department, Department of Endocrinology, Bangladesh Institute of Research and Rehabilitation in Diabetes, Endocrine and Metabolic Disorders
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIRDEM; BADAS-ERC/EC/24/13 (Other: BADAS)
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Type2diabetes
Keywords: Omarigliptin; Type 2 Diabetes Mellitus; DPP-4 inhibitor; Real world evidence; Bangladesh; T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 2-(2,5-difluorophenyl)-5-(2-(methylsulfonyl)-2,6-dihydropyrrolo(3,4-c)pyrazol-5(4H)-yl)tetrahydro-2H-pyran-3-amine; Sulfonylurea Compounds; Metformin; Thiazolidinediones; Glycoside Hydrolase Inhibitors; Glucagon-Like Peptide 1; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- Omarigliptin (Experimental): Arm A will include patients receiving omarigliptin. However, the decision to initiate omarigliptin will be at the treating physician's discretion. The dose of omarigliptin will be 12.5 mg or 25 mg, oral tablet, once weekly decided by the respective physician.
  Interventions: Drug: Omarigliptin
- Sulphonylureas (Active Comparator): This Arm will include patients receiving Sulphonylureas (Gliclazide/ Glipizide/ Glimepiride/ Tolbutamide) according to the physician's choice.
  Interventions: Drug: Sulphonylureas
- Metformin (Active Comparator): This Arm will include patients receiving Metformin according to the physician's choice.
  Interventions: Drug: Metformin
- DPP-4i (Active Comparator): This Arm will include patients receiving DPP-4i other than sitagliptin, vildagliptin, saxagliptin, linagliptin, and alogliptin etc.
  Interventions: Drug: Other DPP4-i
- Thiazolidinediones (Active Comparator): This Arm will include patients receiving Thiazolidinediones (Glitazones, pioglitazone, rosiglitazones)
  Interventions: Drug: Thiazolidinediones
- Alpha-Glucosidase Inhibitor (Active Comparator): This Arm will include patients receiving Alpha-Glucosidase Inhibitor (Acarbose, Miglitol, etc.)
  Interventions: Drug: Alpha-Glucosidase Inhibitor
- Glucagon-Like Peptide-1 (Active Comparator): This Arm will include patients receiving Glucagon-Like Peptide-1
  Interventions: Drug: Glucagon-Like Peptide-1
- Receptor Agonists (GLP1RA) (Active Comparator): This Arm will include patients receiving Exenatide, lixisenatide, liraglutide, albiglutide, dulaglutide, and semaglutide etc.
  Interventions: Drug: Receptor Agonists (GLP1RA)
- SGLT2 inhibitors (Active Comparator): This Arm will include patients receiving Empagliflozin, Ertugliflozin, Canagliflozin, Dapagliflozin
  Interventions: Drug: SGLT2 inhibitors

INTERVENTIONS:
Drug: Omarigliptin — Chemical name: MK-3102 Class: Dipeptidyl peptidase-4 (DPP-4) inhibitor
  Mechanism of Action:
  Inhibits DPP-4 enzyme, thereby increasing incretin levels. Enhances glucose-dependent insulin secretion. Suppresses glucagon secretion. Improves β-cell function of the pancreas. Reduces hepatic glucose output. Administration: Once-weekly oral dosing.
  Arms: Omarigliptin
Drug: Sulphonylureas — Chemical Name: Sulphonylureas Class: Sulphonylureas
  Mechanism of Action:
  Stimulates insulin release from pancreatic beta cells. Enhances the sensitivity of beta cells to glucose. Reduces hepatic glucose production. Increases peripheral glucose uptake and utilization. Administration: Typically administered once or twice daily, depending on the specific medication and patient needs.
  Arms: Sulphonylureas
Drug: Metformin — Chemical Name: Metformin Class: Biguanide
  Mechanism of Action:
  Decreases hepatic glucose production. Improves insulin sensitivity in peripheral tissues. Enhances peripheral glucose uptake and utilization. Reduces intestinal absorption of glucose. Administration: Administered orally, usually once or twice daily with meals.
  Arms: Metformin
Drug: Other DPP4-i — Chemical Names: Sitagliptin, Vildagliptin, Saxagliptin, Linagliptin, Alogliptin Class: Dipeptidyl Peptidase-4 (DPP-4) Inhibitors
  Mechanism of Action:
  Inhibits DPP-4 enzyme, thereby increasing incretin levels. Enhances glucose-dependent insulin secretion. Suppresses glucagon secretion. Improves β-cell function of the pancreas. Reduces hepatic glucose output. Administration: Typically administered orally once daily. Dosage may vary depending on the specific medication and patient needs.
  Arms: DPP-4i
Drug: Thiazolidinediones — Chemical Name: Thiazolidinediones (e.g., Pioglitazone, Rosiglitazone) Class: Thiazolidinediones (TZDs)
  Mechanism of Action:
  Activates peroxisome proliferator-activated receptor-gamma (PPAR-γ) in adipose tissue, muscle, and liver.
  Increases insulin sensitivity in peripheral tissues. Enhances glucose uptake and utilization in muscle and adipose tissue. Reduces hepatic glucose production. Administration: Administered orally, typically once daily. Dosage may vary based on the specific medication and patient response.
  Arms: Thiazolidinediones
Drug: Alpha-Glucosidase Inhibitor — Chemical Name: Alpha-Glucosidase Inhibitors (e.g., Acarbose, Miglitol) Class: Alpha-Glucosidase Inhibitors
  Mechanism of Action:
  Inhibits alpha-glucosidase enzymes in the small intestine. Delays the breakdown and absorption of complex carbohydrates. Reduces postprandial blood glucose levels. Administration: Administered orally, typically taken with the first bite of each main meal. Dosage may vary based on the specific medication and patient response.
  Arms: Alpha-Glucosidase Inhibitor
Drug: Glucagon-Like Peptide-1 — Chemical Name: Glucagon-Like Peptide-1 (GLP-1) Receptor Agonists (e.g., Exenatide, Liraglutide, Dulaglutide, Semaglutide) Class: GLP-1 Receptor Agonists
  Mechanism of Action:
  Mimics the action of endogenous GLP-1. Enhances glucose-dependent insulin secretion. Suppresses glucagon secretion. Slows gastric emptying. Promotes satiety and reduces food intake. Improves β-cell function of the pancreas. Administration: Administered via subcutaneous injection, with frequency varying from twice daily to once weekly, depending on the specific medication.
  Arms: Glucagon-Like Peptide-1
Drug: Receptor Agonists (GLP1RA) — Chemical Name: GLP-1 Receptor Agonists (GLP1RA) (e.g., Exenatide, Liraglutide, Dulaglutide, Semaglutide) Class: Glucagon-Like Peptide-1 Receptor Agonists
  Mechanism of Action:
  Activates GLP-1 receptors. Enhances glucose-dependent insulin secretion. Suppresses glucagon secretion. Slows gastric emptying. Promotes satiety and reduces food intake. Improves β-cell function of the pancreas. Administration: Administered via subcutaneous injection, with frequency varying from twice daily to once weekly, depending on the specific medication.
  Arms: Receptor Agonists (GLP1RA)
Drug: SGLT2 inhibitors — Chemical Name: Sodium-Glucose Co-Transporter-2 (SGLT2) Inhibitors (e.g., Canagliflozin, Dapagliflozin, Empagliflozin, Ertugliflozin) Class: SGLT2 Inhibitors
  Mechanism of Action:
  Inhibits SGLT2 in the proximal renal tubules. Reduces reabsorption of filtered glucose from the renal tubules. Increases urinary glucose excretion. Lowers blood glucose levels independently of insulin. Administration: Administered orally, typically once daily. Dosage may vary based on the specific medication and patient response.
  Arms: SGLT2 inhibitors

SUMMARY:
The study titled "Efficacy and Safety of Omarigliptin, A Weekly Dipeptidyl Peptidase-4 Inhibitor for Type 2 Diabetes Management: Real-World Evaluation in Bangladesh" aims to assess the real-world effectiveness and safety of omarigliptin in managing newly diagnosed type 2 diabetes mellitus (T2DM) patients. Conducted at BIRDEM General Hospital, this 12-month observational study involves 938 patients aged 18 years or older, newly diagnosed with T2DM, with no prior use of antidiabetic medications.

T2DM is a growing global health concern, necessitating effective treatment strategies. Omarigliptin, a once-weekly DPP-4 inhibitor, has shown promising results in clinical trials worldwide. However, its real-world efficacy and safety in diverse populations like Bangladesh remain under-explored. This study aims to fill this gap by evaluating omarigliptin in a typical clinical setting in Bangladesh, potentially providing valuable insights for healthcare providers.

Study Objectives: To assess the real-world efficacy and safety of omarigliptin in managing newly diagnosed T2DM. Specific objectives include evaluating glycemic control (HbA1C levels), safety regarding adverse events, and other outcomes such as changes in fasting plasma glucose, electrolyte levels, liver enzymes, creatinine, and lipid profile.

Methodology: Conducted in the Department of Endocrinology at BIRDEM General Hospital over 12 months, the study population includes newly diagnosed T2DM patients divided into two groups: those receiving omarigliptin and those receiving other antidiabetic agents. Sample size calculation determined 469 patients per group, accounting for a 15% dropout rate.

Inclusion Criteria:

* Newly diagnosed T2DM (according to ADA guidelines) aged ≥ 18 years
* HbA1C levels between ≥7.0% and ≤10.0%
* Stable doses of antidiabetic drugs for at least 4 weeks

Exclusion Criteria:

* Prescribed insulin for diabetes management
* Significant weight loss, hypersensitivity to antidiabetic drugs, type 1 diabetes, ketoacidosis, active liver disease, significant cardiovascular disease, malignancy, hematological disorders, pregnancy, and severe renal impairment, among others.

Study Variables: Data will be collected on demographic variables (age, gender, socio-economic status, BMI), laboratory variables (HbA1C, fasting blood glucose, lipid profile, creatinine, electrolytes, ALT, and postprandial glucose), and adverse events (respiratory infections, headaches, gastrointestinal issues, joint pain).

Study Procedure: Patients will receive personalized antidiabetic treatment with or without omarigliptin, alongside standard dietary and exercise recommendations. Follow-up assessments will occur at 14 days, 3 months, and 6 months post-enrollment. Data will be collected through interviews, physical exams, and laboratory tests, recorded in case record forms (CRFs).

Adverse Event Monitoring: Adverse events (AEs) and serious adverse events (SAEs) will be monitored throughout the study. Participants will be instructed to record any side effects in a treatment diary and contact the study team as needed. AEs include any unfavorable medical occurrences, while SAEs involve life-threatening conditions, hospitalization, or significant disability.

Data Analysis: Data will be analyzed using SPSS Version 23. Descriptive analyses will investigate participant characteristics, with statistical significance set at p < 0.05. Parametric variables will be assessed using Student's t-test, and Spearman's correlation will be used for correlations. Regression analyses will also be performed.

Ethical Considerations: The study will adhere to the Declaration of Helsinki and other ethical guidelines. Approval will be sought from the Institutional Review Board (IRB) of BIRDEM. Written informed consent will be obtained from all participants before enrollment.

DETAILED DESCRIPTION:
IIntroduction Type 2 diabetes mellitus (T2DM) is a chronic metabolic disorder characterized by insulin resistance and impaired insulin secretion, leading to elevated blood glucose levels. Associated with significant morbidity and mortality, T2DM complications include cardiovascular disease, nephropathy, retinopathy, and neuropathy. With its increasing global prevalence, especially in developing countries like Bangladesh, T2DM poses substantial public health challenges.

Management of T2DM requires a combination of lifestyle modifications and pharmacotherapy to achieve and maintain glycemic control. Dipeptidyl peptidase-4 (DPP-4) inhibitors, a class of oral antidiabetic agents, enhance the incretin system, thereby increasing insulin secretion and decreasing glucagon release in a glucose-dependent manner. Omarigliptin, a novel, once-weekly DPP-4 inhibitor, has demonstrated efficacy and safety in clinical trials, but its real-world effectiveness and safety profile, particularly in diverse populations, remain underexplored.

Study Objectives The primary objective of this study is to evaluate the real-world efficacy and safety of omarigliptin in managing newly diagnosed T2DM patients in Bangladesh. Specific objectives include assessing glycemic control (measured by HbA1c levels), monitoring adverse events, analyzing changes in fasting plasma glucose (FPG), postprandial glucose (PPG), and other laboratory parameters, and comparing outcomes with other antidiabetic agents.

Methodology

Study Design:

This is an observational, real-world study conducted over 12 months at the Department of Endocrinology, BIRDEM General Hospital, Dhaka, Bangladesh. The study includes newly diagnosed T2DM patients aged 18 years or older. Participants are divided into two groups: those receiving omarigliptin and those receiving other antidiabetic agents.

Study Population:

Participants will be newly diagnosed T2DM patients attending BIRDEM General Hospital. They will be managed with either omarigliptin or other antidiabetic agents, with personalized treatment regimens decided by the attending physician based on clinical conditions.

Data Collection:

Data will be collected through patient interviews, physical examinations, and laboratory tests. All data will be recorded in standardized case record forms (CRFs). Follow-up assessments will occur at 14 days, 3 months, and 6 months post-enrollment.

Study Variables:

Demographic and laboratory variables will be recorded, including age, gender, socio-economic status, BMI, HbA1c, fasting blood glucose, postprandial glucose, lipid profile, serum creatinine, electrolytes, and liver enzymes. Adverse events will also be tracked and categorized.

Study Procedure:

Participants will receive personalized antidiabetic treatment, including lifestyle modifications and dietary recommendations. The treatment regimen, including the use of omarigliptin, will be determined by the attending physician.

Follow-Up Assessments:

Follow-up assessments will occur at 14 days, 3 months, and 6 months post-enrollment. During these follow-up visits, the following parameters will be checked:

* 14 Days:

  * Review of treatment adherence and any immediate side effects
  * Physical examination
  * Fasting plasma glucose (FPG) levels
  * Recording any adverse events (AEs)
* 3 Months:

  * Physical examination
  * HbA1c levels
  * Fasting plasma glucose (FPG) levels
  * Postprandial glucose (PPG) levels
  * Lipid profile (total cholesterol, LDL, HDL, triglycerides)
  * Serum creatinine
  * Electrolytes
  * Liver enzymes (ALT)
  * Recording any adverse events (AEs)
* 6 Months:

  * Comprehensive physical examination
  * HbA1c levels
  * Fasting plasma glucose (FPG) levels
  * Postprandial glucose (PPG) levels
  * Lipid profile (total cholesterol, LDL, HDL, triglycerides)
  * Serum creatinine
  * Electrolytes
  * Liver enzymes (ALT)
  * Monitoring for serious adverse events (SAEs)
  * Final recording of adverse events (AEs)

Adverse Event Monitoring:

Adverse events (AEs) and serious adverse events (SAEs) will be monitored throughout the study. Participants will record any side effects in a treatment diary and contact the study team as needed. AEs include any unfavorable medical occurrences, while SAEs involve life-threatening conditions, hospitalization, or significant disability.

Data Analysis:

Data will be analyzed using SPSS Version 23. Descriptive statistics will summarize patient characteristics. Paired t-tests will analyze changes in laboratory parameters. Comparisons between groups will be made using Student's t-tests and chi-square tests. Statistical significance is set at p < 0.05. Regression analysis will identify predictors of treatment response.

Ethical Considerations:

The study will adhere to the Declaration of Helsinki and relevant local guidelines. Ethical approval will be obtained from the Institutional Review Board (IRB) of BIRDEM. Written informed consent will be obtained from all participants before enrollment.

Expected Outcomes:

The study aims to provide real-world evidence on the efficacy and safety of omarigliptin in a typical clinical setting. By comparing outcomes with other antidiabetic agents, the study will help elucidate the relative benefits and risks of omarigliptin, aiding healthcare providers in making informed treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed T2DM (according to American Diabetic Association, ADA guideline) aged (≥ 18 years) treated with stable doses of antidiabetic medications (with or without omarigliptin) along with standard diet and exercise
* HbA1C ranged ≥7.0% and ≤10.0%
* Stables doses of drug at least 4 weeks

Exclusion Criteria:

* Newly diagnosed T2DM who will be prescribed insulin for diabetes management
* History of significant weight loss in past 6 months (more than or equal to 5 kg in 1 month)
* Hypersensitivity to any antidiabetic drug
* Type 1 diabetes, a history of ketoacidosis,
* Active liver disease,
* Significant cardiovascular disease,
* A history of malignancy,
* Hematological disorders
* Omarigliptin at any time.
* Any acute condition (acute coronary syndrome, acute stroke etc.)
* Pregnancy and lactation
* eGFR) <30 mL/min/1.73 m2
* ALT (alanine aminotransferase)->2 times the upper limit of the normal
* AST (aspartate aminotransferase)->2 times the upper limit of the normal
* TSH-increased or decreased than the normal range
* Hemoglobin <11 g/dL (male) or <10 g/dL (female),
* Triglycerides >600 mg/dL, or
* C-peptide <0.6 ng/mL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 938 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Glycemic Control as Measured by HbA1c Levels | Baseline assessment. Follow-up visits at 14 days, 3 months, and 6 months post-enrollment.
  Evaluation of the efficacy of omarigliptin in managing glycemic control among newly diagnosed Type 2 Diabetes Mellitus (T2DM) patients in a real-world clinical setting.

CONTACTS AND LOCATIONS:
Overall Officials: Faria Afsana, MD, Principal Investigator — Associate Professor, BIRDEM
Locations (1):
- BIRDEM General Hospital, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided